CLINICAL TRIAL: NCT00853853
Title: Randomized Trial Comparing Standard Ferguson Technique With the EnSeal Device During Hemorrhoidectomy
Brief Title: EnSeal Device Versus Ferguson Technique in Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Steven Schechter, M.D. (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Steven Schechter, M.D., Site Director of Colorectal Fellowship program for The Miriam Hospital affiliated with Brown University Program in Colorectal Surgery, The Miriam Hospital
Organization: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2048-08
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoidectomy; Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. EnSeal Device (Active Comparator): The EnSeal device cuts and seals with heat energy leaving a sutureless wound, which heals with security against bleeding. The device is able to seal blood vessels up to 7mm and hemorrhoidal vessels are much smaller than this size.
  Interventions: Device: EnSeal Device
- 2. Ferguson Hemorrhoidectomy (Active Comparator): The closed Ferguson hemorrhoidectomy technique is a gold standard operation that has been in existence for 50 years. This operation is done under general or intravenous sedation, and the operating surgeon uses a special clamp to go across the hemorrhoidal complex followed by excision of the hemorrhoid. Sutures that dissolve are then placed at the root of the hemorrhoid, securely tied, and then run about the clamp. The clamp is removed and then the suture tightened, then the suture line is reinforced.
  Interventions: Procedure: Ferguson Hemorrhoidectomy technique

INTERVENTIONS:
Device: EnSeal Device — Hemorrhoidectomy using the EnSeal Device, which is an instrument cuts and seals with heat energy leaving a sutureless wound, which heals with security against bleeding.
  Arms: 1. EnSeal Device
Procedure: Ferguson Hemorrhoidectomy technique — The closed Ferguson hemorrhoidectomy technique is a gold standard operation that has been in existence for 50 years. This operation is done under general or intravenous sedation, and the operating surgeon uses a special clamp to go across the hemorrhoidal complex followed by excision of the hemorrhoid. Sutures that dissolve (such as 3.0 vicryl) are then placed at the root of the hemorrhoid, securely tied, and then run about the clamp. The clamp is removed and then the suture tightened, then the suture line is reinforced. This can be done from 1-3 hemorrhoidal groups at a single time.
  Arms: 2. Ferguson Hemorrhoidectomy

SUMMARY:
This study will compare hemorrhoid surgery by comparing a sutureless heating device with the old standard hemorrhoid surgery. Patients will be followed closely for wound healing and satisfaction.

Hypothesis: The sutureless device will be less painful for the patient and easier for the surgeon to perform.

DETAILED DESCRIPTION:
The EnSeal Device is approved for laparoscopic surgery in ligating and dividing vascular tissue during abdominal surgery. Electrical energy is converted into heat energy and resultant simultaneous division of tissues. This allows surgery to be bloodless and sutureless. This device is being used in the current study in the treatment of hemorrhoidal disease where vascular tissue is excised in bloodless and sutureless fashion. The device is FDA-approved for laparoscopic surgery. This is currently being used in institutions throughout the United States and Europe.

This study is looking at the EnSeal device and comparing it to a gold standard hemorrhoidal procedure to see if the OR procedure can be simplified and the postoperative course improved.

The trial is a randomized, controlled, prospective study. Patients will be informed of the two techniques being studied and will be randomized in the operating room by opening up an envelope with the procedure to be employed inside. The envelopes will be numbered 1 through 100, with 50 envelopes containing a slip of paper stating that the surgery will be done using the Ferguson technique and 50 envelopes containing a slip of paper stating the that the surgery will be done using the EnSeal device. These slips of paper will be placed in the envelopes and sealed. The envelopes will be mixed up by someone not involved in the study and then numbered 1 through 100. No one will know which surgical technique will be used on the patient until the surgeon opens the envelope on the day of surgery.

Patients will be followed postoperatively in the office during week 1, week 4, and week 12. At this time, they will be assessed for postoperative complications including but not limited to: bleeding, urinary retention, infection, fecal impaction, hospital re-admission and pain. Delayed complications will also be followed including urinary retention, impaired healing, constipation, abscess, fistula formation, fissure, stenosis, fecal incontinence, and flatus incontinence. The patient's pain score will be assessed using the Universal Pain Assessment Tool, allowing the patient to describe their pain level on a scale between 1 and 10.

ELIGIBILITY:
Inclusion Criteria:

1. Men & woman between ages 18-80.
2. ASA level I, II, and III.
3. External hemorrhoids may or may not be present.
4. Internal hemorrhoids at least Grade II, III, and IV.

Exclusion Criteria:

1. Age less than 18, or greater than 80.
2. ASA level IV.
3. Grade I internal hemorrhoids.
4. Patients on Coumadin, Plavix, or other anticoagulant.
5. Associated procedure such as sphincterotomy, drainage of abscess, fistulotomy, or the like.
6. Pregnancy - Women who have a positive urine pregnancy test pre-op will be excluded from the study.
7. Inflammatory bowel disease.
8. History of chronic active hepatitis B, C, or HIV infection.
9. Lactating women.
10. Inability to follow up with surgeon in office at 1 week, 4 weeks, and 3 months postoperatively.
11. Prior chronic narcotic use (> 30 days)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
to examine the advantage and disadvantages of the EnSeal device as it applies to hemorrhoidal surgery and document outcomes as compared to the traditional closed Ferguson hemorrhoidectomy | 1 week, 4 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schechter, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States